CLINICAL TRIAL: NCT04158297
Title: Extracorporeal Shock Wave Lithotripsy Versus Single Operator Pancreatoscopy and Intraductal Lithotripsy for the Treatment of Pancreatic Duct Stones
Brief Title: ESWL Versus SOPIL for Treatment of Pancreatic Duct Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jeffrey Easler, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1909140534
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pancreatitis; Pancreatic Duct Stone
Keywords: Extracorporeal shock wave lithotripsy; Intraductal lithotripsy
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESWL (Active Comparator): Extracorporeal shock wave lithotripsy for the treatment of pancreatic duct stones
  Interventions: Procedure: ESWL vs SOPIL
- SOPIL (Active Comparator): Single Operator Pancreatoscopy and intraductal lithotripsy for the treatment of pancreatic duct stones
  Interventions: Procedure: ESWL vs SOPIL

INTERVENTIONS:
Procedure: ESWL vs SOPIL — To compare the efficacy of single operator pancreatoscopy (SOP) with intracorporeal lithotripsy (SOPIL) to extracorporeal shock wave lithotripsy (ESWL) for the treatment of main pancreatic duct stones (MPDS) in patients with chronic pancreatitis.

SUMMARY:
Pancreatic duct stones can cause obstruction of the main pancreatic duct leading to abdominal pain, exocrine pancreatic insufficiency, and recurrent acute pancreatitis. By removing pancreatic duct stones, the obstruction can be relieved, and this can improve symptoms. Small stones can be removed with standard endoscopic retrograde cholangiopancreatography (ERCP) and stone removal, but larger stones may require lithotripsy to break up the stone before removal. The two current methods of lithotripsy include extracorporeal shock wave lithotripsy (ESWL) and single operator pancreatoscopy with intracorporeal lithotripsy (SOPIL).

ESWL is based on concentrating shock wave energy to the stone through an external device. SOPIL is a newer technique based on direct visualization of the stone during ERCP and targeting the stone with a shock wave catheter. There are currently no studies directly comparing ESWL to SOPIL for breaking apart stones in the pancreatic duct, so this study is designed to compare the two techniques.

Objective #1: Obtain pilot data to determine the optimal method of clearing large MPDS Objective #2: Obtain pilot data to assess how effective large MPDS clearance is in improving long term patient centered outcomes Objective #3: Obtain pilot data to measure the cost effectiveness of large MPDS clearance

ELIGIBILITY:
Inclusion Criteria:

* MPDS located in the head, neck, or neck/body junction of the pancreas
* MPDS > 5 mm in size
* Abdominal CT scan, Endoscopic ultrasound, or prior ERCP demonstrating MPDS
* Abdominal pain related to MPDS
* Previously failed ERCP performed with intent to clear MPDS, OR MPDS determined by treating physicians to not be amenable to clearance by standard ERCP techniques

Exclusion Criteria:

* MPDS predominantly located in the body and tail of pancreas
* Any obstructing MPDS > 5 mm located in the body and tail of pancreas
* Known pancreatic head stricture precluding passage of the pancreatoscope with endoscopic stone extraction based on prior imaging or prior ERCP
* Pancreatic head mass
* Impacted MPDS located at the pancreatic duct orifice
* Prior attempts at ESWL or SOPIL for MPDS
* Walled off pancreatic necrosis
* Active alcohol use, defined as any alcohol use within 2 months
* Surgically altered anatomy (see text)
* Gastric outlet obstruction or obstruction precluding passage of the endoscope
* Standard contraindications to ERCP
* Implanted cardiac pacemakers or defibrillators
* Known calcified aneurysms in the path of the shockwave
* Age < 18 years, pregnancy, incarceration, unwillingness/inability to provide informed consent, or anticipated inability to follow protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Technical success of complete or partial clearance (≥80% stone clearance) of large main pancreatic duct stone | Up to 24 weeks
  This will be described as a proportion of patients with stone clearance. This is defined by the endoscopist's interpretation of the pancreatogram during the time of ERCP and/or subsequent imaging studies. Two blinded endoscopists will review the final pancreatogram to confirm clearance of MPDS
Mean number of lithotripsy and ERCP procedures needed for clearance of stones or in the attempt to clear stones | Up to 24 weeks
  Combined lithotripsy and ERCP procedures
Procedural related adverse events | Up to 24 weeks
  This will be described as a proportion of patients who develop post-procedure pancreatitis, bleeding, infection, perforation, organ injury, symptomatic hematoma, or Steinstrasse resulting in acute stone impaction at the papilla

SECONDARY OUTCOMES:
Change in pain scores | through study completion, an average of 1 year
  Change in Izbicki pain scores from baseline at 3 months, 6 months, 9 months, and 12 months. The Izbicki pain scale is a validated pain score for chronic pancreatitis using a visual analog scale, frequency of pain, requirement of pain medication, and pain affecting functional ability. The score ranges from 0 to 100 with higher scores suggesting more pain.
Change in quality of life based on chronic pancreatitis specific instruments: PANQOLI | through study completion, an average of 1 year
  Change in the pancreatitis quality of life instrument (PANQOLI) scores from baseline at 3 months, 6 months, 9 months, and 12 months. The PANQOLI score is a validated quality of life score for chronic pancreatitis with specific focus on the domains of physical function, role function, emotional function, and self-worth. The score ranges from 11 to 103, which higher scores suggesting better quality of life.
Change in narcotic pain medication usage | through study completion, an average of 1 year
  Change in daily morphine milligram equivalent usage from baseline at 3 months, 6 months, 9 months, and 12 months
Change in exocrine insufficiency | through study completion, an average of 1 year
  This will be described as a proportion of patients who experience weight gain, resolution of steatorrhea, or no longer require pancreatic enzyme supplementation after stone clearance at 3 months, 6 months, 9 months, and 12 months

OTHER OUTCOMES:
Mean cost of care for stone clearance | up to 24 weeks
  Costs will be estimated by procedural fees including the cost of ESWL, lithotripsy, ERCP, anesthesia, and fluoroscopy.
Health care utilization | through study completion, an average of 1 year
  Change in frequency of emergency room visits or hospitalization after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery J Easler, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No